CLINICAL TRIAL: NCT06270992
Title: Developing an Artificial Intelligence-based Diagnostic Method Based on Oral Microbiome for Non-invasive Diagnosis of Lung Cancer
Brief Title: Oral Microbiome Diagnostics of Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aycan Gundogdu, Associate Professor, TC Erciyes University
Other Study IDs: 123R030
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: oral microbiome; non-invasive diagnosis; artificial intelligence
MeSH Terms: conditions — Lung Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Oral swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung cancer group: 192 patients diagnosed with lung cancer with the following inclusion criteria:
  * To be between the ages of 18 and 65,
  * Not having been previously diagnosed with and treated for lung cancer,
  * Not having received any cancer treatment in the last 2 years,
  * Not having been operated on within the last two years,
  * Not having a hospitalization history in the last year,
  * Not having used antibiotics in the last six months,
  * Not having used products manufactured to support the oral microbiome, such as probiotic (lozenges, sublingual drops) for at least the last six months,
  * Not being pregnant, not breastfeeding,
  * Not having undergone dental procedures such as root canal treatment, implants, prostheses, tooth extraction, fillings in the last 6 months, Not having dominant immune-origin lesions , viral-origin lesions, dominant bacterial infections like tonsillitis, and/or thermal or chemical mucosal traumas in the mouth.
  Interventions: Diagnostic Test: NCCN (National Comprehensive Cancer Network) diagnosis
- Benign lung disease group: 192 patients diagnosed with non-cancer diseases with the following inclusion criteria:
  * To be between the ages of 18 and 65,
  * To have visited our clinic with complaints related to the lungs and/or respiratory tract,
  * Not having been diagnosed with lung cancer after clinical evaluation,
  * Not having received any cancer treatment in the last 2 years,
  * Not having been operated on within the last two years,
  * Not having a hospitalization history in the last year,
  * Not having used antibiotics in the last six months,
  * Not having used products manufactured to support the oral microbiome, such as probiotics for at least the last six months,
  * Not being pregnant or breastfeeding,
  * Not having undergone dental procedures such as root canal treatment, implants, prostheses, tooth extraction, fillings in the last 6 months,
  * Not having dominant immune-origin lesions, viral-origin lesions, dominant bacterial infections like tonsillitis, and/or thermal or chemical mucosal traumas in the mouth.
  Interventions: Diagnostic Test: NCCN (National Comprehensive Cancer Network) diagnosis
- Healthy control group: 292 individuals without lung cancer or another lung disease diagnosis with the following inclusion criteria:
  * To be between the ages of 18 and 65,
  * Not to have a diagnosed lung disease or suspicion thereof,
  * Not to have complaints related to the lungs and/or respiratory tract,
  * Not to have alcohol or severe substance dependency,
  * Not having a hospitalization history in the last year,
  * Not having used antibiotics in the last six months,
  * Not having used products manufactured to support the oral microbiome, such as probiotics (lozenges, sublingual drops) for at least the last six months,
  * Not being pregnant or breastfeeding,
  * Not having undergone dental procedures such as root canal treatment, implants, prostheses, tooth extraction, fillings in the last 6 months,
  * Not having dominant immune-origin lesions, viral-origin lesions, dominant bacterial infections like tonsillitis, and/or thermal or chemical mucosal traumas in the mouth.

INTERVENTIONS:
Diagnostic Test: NCCN (National Comprehensive Cancer Network) diagnosis — For diagnostic evaluation, the necessary procedures from the standard protocols consisting of anamnesis, physical examination, laboratory tests, radiological imaging methods, and tissue biopsy will be followed. Computerized Tomography (CT) and Positron Emission Tomography-Computed Tomography (PET-CT) will be used as imaging methods, while fiberoptic bronchoscopy and video-assisted mediastinoscopy will be applied for tissue diagnosis and staging.
  Groups: Benign lung disease group; Lung cancer group

SUMMARY:
The study aims to develop a deep learning-based diagnostic method for lung cancer using the oral microbiome. This innovative approach involves establishing an observational cohort of 576 individuals, including lung cancer patients, non-cancerous benign lung disease patients, and healthy controls, to collect tongue swab samples for 16S rRNA sequencing. Additionally, an international cohort of approximately 1700 individuals will be formed using in silico data. The project will utilize deep learning methods to analyze all data integratively and develop an AI diagnostic algorithm capable of distinguishing lung cancer patients from others. The diagnostic method's performance will be tested in a pilot clinical trial with 96 individuals using a PRoBE design. Led by experts in chest surgery, molecular microbiology, and bioinformatics, the project spans over 30 months and aims to create a non-invasive, easily accessible lung cancer screening method that could lead to significant diagnostic advancements and potential spin-off companies in the field of liquid biopsy/molecular diagnosis.

DETAILED DESCRIPTION:
Cancer is a global health issue that is on an increasing trend in terms of incidence and mortality rates, hindering the increase in life expectancy. According to the World Health Organization, lung, colorectal, and liver cancers are among the most common causes of cancer-related deaths. In Turkey, the incidence and mortality rates of lung cancer are higher than the world average. are among the risk factors that may increase the risk of lung cancer. In addition to risk factors like family history, smoking, different studies have shown that dysbiotic oral microbiome may contribute to the risk of lung cancer.

The oral microbiome is the second most diverse microenvironment in our body and has been associated with many diseases, including lung cancer. Studies to date on lung cancer-oral microbiome have generally involved designs aimed at resolving cause-and-effect relationships through statistical differences and/or mechanisms involving microbiome units.

However, there is no literature on any study aimed at developing a deep learning-based diagnostic method that focuses on the oral microbiome.Therefore, the proposed study aims to develop a microbiome based deep learning diagnostic method for lung cancer diagnosis. To this end, an observation cohort will be established consisting of 192 lung cancer patients, 192 non-cancerous benign lung disease patients, and 192 healthy controls. Tongue swab samples belonging to the cohort will be collected, and 16S rRNA sequencing will be performed. At the same time, an international observation cohort of approximately 1700 individuals will be created using in silico data. All data will be analyzed integratively, and an artificial intelligence diagnostic algorithm that can differentiate lung cancer patients from other lung diseases and healthy individuals will be developed using deep learning methods. In the final stage, the performance of the diagnostic method developed for a pilot clinical trial cohort of 96 individuals will be tested using a PRoBE (prospective specimen collection before outcome ascertainment and retrospective blinded evaluation) design.

The original aspects of the project are the proposal of a novel design in the literature, the creation of an experimental design/clinical trial and the presentation of a potential solution proposal that may have a high impact on an important diagnostic problem.

If the project is successfully completed, an artificial intelligence-based method that can potentially diagnose lung cancer through non-invasive oral microbiome samples will be developed. In addition to its patentability, if the method is further developed (in the medium to long term) into a product, it will enable lung cancer screening to be easily performed even in primary healthcare institutions with a simple oral swab sample.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18 and 65,
* Not to have a diagnosed lung disease or suspicion thereof,
* Not to have complaints related to the lungs and/or respiratory tract,
* Not to have alcohol or severe substance dependency,
* Not having a hospitalization history in the last year,
* Not having used antibiotics in the last six months,
* Not having used products manufactured to support the oral microbiome, such as probiotics (lozenges, sublingual drops) for at least the last six months,
* Not being pregnant or breastfeeding,
* Not having undergone dental procedures such as root canal treatment, implants, prostheses, tooth extraction, fillings in the last 6 months
* Not having dominant immune-origin lesions (such as aphthous ulcers, erythema multiforme, pemphigus), viral-origin lesions (such as herpes, Koplik spots, herpangina), dominant bacterial infections like tonsillitis, and/or thermal or chemical mucosal traumas in the mouth.

Exclusion Criteria:

* Not to satisfy inclusion or declining to participate even though all the inclusion criteria are satisfied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population consists of a lung cancer group of 192 patients, a non-lung cancer benign lung disease group of 192 patients, and 292 healthy controls. Each subgroups are gender and age matched.
Sampling Method: Non-Probability Sample
Enrollment: 676 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostics accuracy assessment | 30 months
  Diagnostic technology under investigation will be evaluated using sensitivity, specificity, area under receiver operating curve. Cross validation will be used for testing and NCCN diagnosis and patient follow-ups will be considered as the ground truth.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR